CLINICAL TRIAL: NCT00321100
Title: Phase II Study of the Combination of Cetuximab, Capecitabine, and Oxaliplatin With Out Without Bevacizumab as Initial Therapy for Metastatic Colorectal Cancer
Brief Title: Combination of Cetuximab, Capecitabine, and Oxaliplatin With or Without Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment closed 10/15/2008 based on data about KRAS.
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-GI-002
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Neoplasms
Keywords: metastatic; colorectal; cancer; initial therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Bevacizumab; Cetuximab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab (Active Comparator): Cetuximab 400 mg/m2 IV initial dose (cycle 1 day 1 only), then 250mg/m2 IV weekly of each 21 day cycle; Oxaliplatin 130mg/m2 IV day 1 of each 21 day cycle; Capecitabine 850mg/m2 PO every 12 hours days 1-14 of each 21 day cycle; Bevacizumab 7.5mg/kg IV day 1 of each 21 day cycle
  Interventions: Drug: bevacizumab; Drug: cetuximab; Drug: Oxaliplatin; Drug: Capecitabine
- Cetuximab, Oxaliplatin, Capecitabine (Active Comparator): Cetuximab 400 mg/m2 IV initial dose (cycle 1 day 1 only), then 250mg/m2 IV weekly of each 21 day cycle; Oxaliplatin 130mg/m2 IV day 1 of each 21 day cycle; Capecitabine 850mg/m2 PO every 12 hours days 1-14 of each 21 day cycle
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: bevacizumab — Bevacizumab 7.5mg/kg IV day 1 of each 21 day cycle
  Other Names: Avastin
  Arms: Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab
Drug: cetuximab — Cetuximab 400mg/m2 IV initial dose (cycle 1 day 1 only), then 250mg/m2 IV weekly each 21 day cycle
  Other Names: Erbitux
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 IV day 1 every 21 days
  Other Names: Eloxatin
  Arms: Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab
Drug: Capecitabine — Capecitabine 850mg/m2 PO every 12 hours days 1-14 of each 21 day cycle
  Other Names: Xeloda
  Arms: Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab

SUMMARY:
The purpose of this study is to determine the objective response rate of patients with previously untreated metastatic colorectal cancer treated with the combination of cetuximab, capecitabine, and oxaliplatin with out without bevacizumab.

DETAILED DESCRIPTION:
Research has shown that the more drug treatments patients with cancer of the colon or rectum receive, the longer they live. One uses the drugs capecitabine and oxaliplatin which all patients on this study will receive. Bevacizumab is an antibody which blocks blood flow to tumors and increases how long patients with colorectal cancer live. However, it can increase the risk of stroke and heart attack. Bevacizumab is currently a standard part of treatment for colorectal cancer. Cetuximab is an antibody which blocks a protein called EGFR which shrinks colorectal cancer. It may be helpful with initial chemotherapy and with bevacizumab. One goal of this study is to find out the response rate (chance of tumor shrinking) with two treatments for colorectal cancer. All patients will get capecitabine, oxaliplatin and cetuximab. Half will receive bevacizumab. All drugs in this study are approved to treat colorectal cancer. This research study is being done to find the best, safest way to combine these therapies.

ELIGIBILITY:
Inclusion Criteria:

* measurable metastatic adenocarcinoma of the colon or rectum
* no prior systemic therapy for metastatic disease
* adjuvant therapy must have been completed >/=12 months prior to recurrence, prior radiotherapy permitted but must have been completed > 6 months prior to study entry
* must have tumor tissue available for EGFR and thymidine phosphorylase evaluation
* ECOG PS 0-1
* age >/= 18
* adequate organ function: WBC>/=3,000, ANC >/=1,500, platelets>/= 100,000, total bilirubin </= 1.5X ULN, AST&ALT </= 2.5X ULN, create clearance >/= 50mL/min
* negative pregnancy test w/in 72 hours of treatment for women of child bearing potential
* ability to understand and willing to sign written ICF
* able to swallow and absorb oral medication

Exclusion Criteria:

* medical or psychiatric condition which would potentially pose risk to patient by participation (i.e. but not limited to:uncontrolled hypertension, MI w/in 6 months,CNS disease, pregnancy or nursing)
* history of neoplasm (other than non-metastatic skin cancer or carcinoma in situ of cervix) w/in 5 years
* surgical procedure (not including closed biopsy or access port placement), open biopsy, significant traumatic injury w/in 28 days of registration or anticipation of need for surgical procedure while on study, fine needle aspiration or core biopsy w/in 7 days of registration
* urine protein:creatinine ration >/=1.0 at screening
* evidence of bleeding diathesis or coagulopathy (in absence of anticoagulation)
* prior severe infusion reaction to MAB or allergic reaction to capecitabine or oxaliplatin
* underlying neuropathy >/= grade 2
* TIA or CVA w/in 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-04-12; Primary Completion 2009-04 (Actual); Study Completion 2013-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Dotan E, Meropol NJ, Burtness B, Denlinger CS, Lee J, Mintzer D, Zhu F, Ruth K, Tuttle H, Sylvester J, Cohen SJ. A phase II study of capecitabine, oxaliplatin, and cetuximab with or without bevacizumab as frontline therapy for metastatic colorectal cancer. A Fox Chase extramural research study. J Gastrointest Cancer. 2012 Dec;43(4):562-9. doi: 10.1007/s12029-012-9368-3. PMID 22294255

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab: Cetuximab: 400 mg/m2 initial dose (cycle 1 day 1 only), then 250mg/m2 IV weekly of each 21 day cycle
  Oxaliplatin: 130mg/m2 IV day 1 of each 21 day cycle
  Capecitabine: 850mg/m2 PO every 12 hours days 1-14 of each 21 day cycle
  Bevacizumab: 7.5mg/kg IV day 1 of each 21 day cycle
- Cetuximab, Oxaliplatin, Capecitabine: Cetuximab: 400 mg/m2 initial dose (cycle 1 day 1 only), then 250mg/m2 IV weekly of each 21 day cycle
  Oxaliplatin: 130mg/m2 IV day 1 of each 21 day cycle
  Capecitabine: 850mg/m2 PO every 12 hours days 1-14 of each 21 day cycle
Period: Overall Study
Arm/Group | Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab | Cetuximab, Oxaliplatin, Capecitabine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab | Cetuximab, Oxaliplatin, Capecitabine | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 78] | 58 [42 to 74] | 59 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate calculated by the proportion of overall response: CR+PR. Patients were categorized by one of the following (1-4 per RECISTv1.0 criteria on CT, MRI, x-ray; 4-9 considered failure to respond/disease progression):
  1. complete response (CR): Disappearance of all lesions
  2. partial response (PR): >=30% decrease in the sum of the longest diameter of target lesions (SoL); from baseline SoL
  3. stable disease (SD): Neither PR, PD, or CR
  4. progressive disease (PD): >=20% increase in the SoL; from smallest SoL. Or appearance of new lesion
  5. early death from malignant disease
  6. early death from toxicity
  7. early death from other cause
  9) unknown (not assessable, insufficient data)
Time Frame: every 6-9 weeks; from date of first study drug dose until off treatment date (median of 8 cycles; range <1-19)
Population: One patient in Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab Arm was not evaluable for response due to patient discontinuing after experiencing a hypersensitivity reaction to cetuximab during the first treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab | Cetuximab, Oxaliplatin, Capecitabine
Number analyzed (Participants) | 11 | 11
Participants
  Overall response | 4 | 8
  Complete response | 1 | 1
  Partial response | 3 | 7
  Stable disease | 7 | 3

2. Secondary Outcome: Time to Progression (TTP)
Description: Per Response Evaluation Criteria In Solid Tumors (RECISTv1.0) assessed by CT, MRI, x-ray scan:
  Complete response (CR): Disappearance of all lesions Partial response (PR): >=30% decrease in the sum of the longest diameter of target lesions (SoL); from baseline SoL Stable disease (SD): Neither PR, PD, or CR Progressive disease (PD): >=20% increase in the SoL; from smallest SoL. Or appearance of new lesion
Time Frame: every 6-9 weeks; from dose of first study drug to event
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab | Cetuximab, Oxaliplatin, Capecitabine
Number analyzed (Participants) | 11 | 11
months | 8.7 [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported. | 14.4 [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.

3. Secondary Outcome: Overall Survival
Description: Follow-up for survival to be done at 3 month intervals for 2 years, then 6 month intervals for up to 5 years from study registration
Time Frame: From dose of first study drug to last timepoint known to be alive (median follow-up for all patients was 25.9 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab | Cetuximab, Oxaliplatin, Capecitabine
Number analyzed (Participants) | 11 | 11
months | 18 [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported. | 42.5 [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.

ADVERSE EVENTS:
Arm/Group | Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab | Cetuximab, Oxaliplatin, Capecitabine
All-Cause Mortality (participants affected / at risk) | 11/12 | 10/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab, Oxaliplatin, Capecitabine, Bevacizumab (N=12) | Cetuximab, Oxaliplatin, Capecitabine (N=11)
Hypersensitivity reaction (Immune system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 6
Infection with neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 7
Hemmorhage (Vascular disorders) | 6 | 4
DVT (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 6 | 2
Edema (General disorders) | 2 | 1
Fatigue (General disorders) | 11 | 11
Pain (General disorders) | 9 | 9
Fever (General disorders) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry/cracked skin (Skin and subcutaneous tissue disorders) | 3 | 4
Fissures (Skin and subcutaneous tissue disorders) | 7 | 3
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 3
Paronychia (Skin and subcutaneous tissue disorders) | 5 | 7
Rash (Skin and subcutaneous tissue disorders) | 11 | 11
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 7 | 6
Diarrhea (Gastrointestinal disorders) | 9 | 11
Nausea (Gastrointestinal disorders) | 9 | 7
Vomiting (Gastrointestinal disorders) | 5 | 2
Weight loss (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Parasthesias (Nervous system disorders) | 8 | 8
Parasthesias/pain (Nervous system disorders) | 1 | 1
Sensory neuropathy (Nervous system disorders) | 5 | 6
Insomnia (Nervous system disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes